CLINICAL TRIAL: NCT02079454
Title: Valeur Predictive de l'INVOS Sur l'Outcome Cardiaque en Post-opératoire. (French Title)
Brief Title: Post-operative Cardiac Outcome of Non-cardiac Surgery Predicted by INVOS
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: invos0001
Record Dates: First submitted 2011-07-20; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Invos; Peri-operative; Cardiac Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples for troponin I measurement
Oversight: Data Monitoring Committee: No

SUMMARY:
Research aimed to find a correlation with an invos drop and cardiac events in the peri-operative period of non cardiac surgery.

The investigators postulate that a drop in the Invos numbers (with or without significant drop in BP) is associated with a variable degree of cardiac suffering.

The idea is to prevent per and foremostpost-operative myocardial necrosis complications by acting as soon as we have an INVOS drop during anesthesia.

The "cardiac events" will be monitored and defined according to the EHA (european heart association) guidelines.

(Changes of the EKG and/or troponin I values above the threshold). Patient will be monitored per and post operatively.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age minimum 18 years old

Exclusion Criteria:

* Chronic renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with high cardiac comorbidities undergoing a general anesthesia for a surgery of over two hours with bleding potential.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
A composite measurement of major vascular events in the post-operative period | 96 hours post-operative
  Myocardial infarction (measured by positivation of troponin I assay above the defined threshold) associated with clinical data (pain, dyspnea,...) or ST modification on the EKG or apparition of a new LBBB, or new wall abnormalities on the TTE.
  Or new TIAs or CVAs

CONTACTS AND LOCATIONS:
Locations (1):
- cliniques universitaires St Luc, Brussels, Brabant, Belgium